CLINICAL TRIAL: NCT04356664
Title: Benefit of Gonadotropin-releasing Hormone (GnRH) Agonist Before Frozen Embryo Transfer in Patients With Endometriosis and / or Adenomyosis: Randomized Prospective Study
Brief Title: Benefit of GnRH Agonist Before Frozen Embryo Transfer in Patients With Endometriosis and/or Adenomyosis
Acronym: DECATEC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019_0012
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis; Adenomyosis; Infertility, Female
MeSH Terms: conditions — Endometriosis; Adenomyosis; Infertility, Female | interventions — Gonadotropin-Releasing Hormone; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frozen embryo transfer with Hormonal Replacement Therapy (HRT) (No Intervention): Patient will received usual Hormonal Replacement Therapy for a Frozen embryo transfer composed of estrogens and progestins.
- Frozen embryo transfer with HRT and GnRH agonist (Experimental): Patient will received 1 or 2 injection of GnRH agonist priori to usual Hormonal Replacement Therapy for a Frozen embryo transfer composed of estrogens and progestins.
  Interventions: Drug: GnRH agonist

INTERVENTIONS:
Drug: GnRH agonist — One or two intramuscular injections of Decapeptyl 3 mg
  Other Names: Decapeptyl 3 mg
  Arms: Frozen embryo transfer with HRT and GnRH agonist

SUMMARY:
Women suffering from endometriosis and/or adenomyosis may also suffer from infertility. GnRH agonist injection could improve implantation and therefore increase the pregnancy rate in these patients. This study was designed to evaluate effects of the additional of GnRH agonist (single or 2 doses) to the routine oestrogens and progestins use as support before Frozen Embryon Transfer as compared to oestrogens and progestins only.

DETAILED DESCRIPTION:
Endometriosis reveals the presence of glands or endometrial stroma outside the uterus, responsible for pain and infertility. Adenomyosis illustrates an invagination of endometrial islets within the myometrium, leading to a disturbance of its contractile activity, also potentiated by local hyperestrogenism.

These two pathologies are often associated, and express an alteration of the eutopic endometrium by pro-inflammatory markers responsible for a lower implantation rate.

GnRH agonists are known to decrease these pro-inflammatory markers (cytochrome P450 and Cox 2 aromatase) in the eutopic endometrium of women with endometriosis or adenomyosis.

Patients will received 1 or 2 injection of GnRH delay agonist (Decapeptyl 3mg) approximately 1 month before the frozen embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 36 years (women ≥18 years to <36 years) with endometriosis and / or adenomyosis
* Having benefited from In vitro fertilisation /intracytoplasmic micro-injection with freeze all and for whom the frozen embryon transfer of a blastocyst is planned
* A normal uterine cavity
* An MRI showing endometriosis and / or adenomyosis during the inclusion visit
* Having signed a consent form
* Being affiliated to a Health Insurance Plan.

Exclusion Criteria:

* Patient aged <18 years and ≥ 36 years
* BMI> 35
* History of implantation failures (≥ 2)
* Endometrial alterations: synechiae, polyps, myomas, hyperplasia, hematometra
* known hydrosalpinx uni or bilateral
* MRI showing no endometriosis or adenomyosis
* Hypersensitivity to GnRH, GnRH analogues, or any of the excipients of Decapeptyl 3 mg
* Known hypersensitivity to estradiol
* Known hypersensitivity to progesterone
* Known hypersensitivity to acetylsalicylic acid or other nonsteroidal anti-inflammatory drugs
* Known hypersensitivity to folic acid
* Known hypersensitivity to cefixime or an antibiotic in the cephalosporin group
* Known hypersensitivity to levofloxacin or any other quinolone
* History of tendinopathies related to the administration of fluoroquinolones
* Epilepsy
* Hypersensitivity to contrast agents for MRI
* Known or suspected breast cancer or history of breast cancer
* Known or suspected genital tract cancer or history of genital cancer
* known or suspected estrogen-dependent malignant neoplasms
* Undiagnosed genital haemorrhage
* Untreated endometrial hyperplasia
* History of idiopathic venous thrombo-embolic accident or evolving venous thrombo-embolic event (deep vein thrombosis, pulmonary embolism)
* Recent or evolving arterial thromboembolic stroke (eg angina, myocardial infarction)
* Acute liver disease or history of liver disease, until hepatic tests are normalized
* Severe renal insufficiency
* Severe, uncontrolled heart failure
* Evolutionary gastroduodenal ulcer
* History of asthma caused by the administration of salicylates or substances of similar activity, especially nonsteroidal anti-inflammatory drugs
* GnRH Agonist Decapeptyl administered within 6 months prior to transfer
* To be deprived of liberty or under guardianship
* Pregnancy and breast feeding.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Treatment of female infertility
Enrollment: 180 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate in both groups at last visit ultrasound | 3 months after frozen embryon transfer
  Clinical pregnancy will be defined by any cardiac activity detected during the ultrasound performed at the last visit.

SECONDARY OUTCOMES:
Successful implantation rate on the number of patients included | 3 months after frozen embryon transfer
  The implantation rate will be evaluated by the number of successful implantations out of the total number of attempts.
Rates of miscarriages on the number of patients included | 3 months after frozen embryon transfer
  The miscarriage rate will be determined by the number of effective miscarriages over the number of successful implantations.
Side effects related to treatment with Decapeptyl 3 mg | 15 months
  Collection of side effects related to treatment with Decapeptyl 3 mg

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pirtea, Dr, Study Director — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No